CLINICAL TRIAL: NCT06144528
Title: Exploring Imitative Abilities and Stereotypies: Comparing Robots and Human Operators in Autistic Children
Brief Title: Comparing Imitation and Stereotyped Behaviors in Autistic Children: Robots vs. Human Operators
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: CNR-IRIB-PRO-2023-005
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Autism; social robot; imitation; Stereotypies
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Stereotypic Movement Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with autism spectrum condition: Thirty Autism Spectrum Disorder (ASD) children with medium-high functioning, aged 4 to 13 years, IQ > 75, in the absence of motor deficits due to another clinical condition.
  Interventions: Other: QT robot

INTERVENTIONS:
Other: QT robot — In a single session each child will be video-recorded while performing the task. The participant subjects will perform the same task at two different times, once with the human operator and once with the Qt robot. Both tasks will have a duration of approximately 4 minutes. During the first minute, both the operator and the Qt will introduce themselves and ask four questions to the child to deepen the acquaintance. In the second minute, the operator/Qt will tell a story. In the third minute, the operator/Qt will ask to imitate 4 motor movements, while in the fourth minute, the operator/Qt will ask to imitate 4 facial expressions.

SUMMARY:
Virtual QT is a social robot designed to interact with humans in social and educational contexts. Equipped with visual and vocal interfaces, the robot can recognize and respond to various human inputs, providing emotional support and social interaction.

It uses facial expressions, gestures, and movements to communicate, encouraging engagement and supporting learning through playful and educational activities. Its ergonomic design and interactive approach make it suitable for both clinical and educational settings.

The aim of this study is to examine the effectiveness of the QTrobot in interventions for children with Autism Spectrum Disorder (ASD) and to assess whether children's attention and imitation are equally effective with the QTrobot compared to interacting with a human being.

Furthermore, the presence of significant differences between motor and expressive imitation, when interacting with the robot as opposed to a human interlocutor, will be investigated. A key aspect of this investigation is to assess whether the presence of the QTrobot can positively influence the repetitive or stereotyped behaviors exhibited by the children, compared to interaction with a person. Additionally, to further understanding, the children's heart rate will be monitored through the use of a sensor that will allow to evaluate how heart rate affects performance outcomes during interaction with the QTrobot and with a human being.

In this study, children will be recruited to take part in two separate sessions, both involving the same task. During the first session, the task will be carried out between the child and the human operator. Subsequently, in the same task, the child will interact with the QT robot. Throughout both task administrations, the child will wear a sensor to detect their heart rate. Furthermore, all task sessions will be video-recorded to conduct subsequent video analysis and make notes on imitation behaviors and stereotypical actions relevant to the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism
* QI ≥ 75

Exclusion Criteria:

* Motor deficits due to another clinical condition

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Thirty children with Autism Spectrum Disorder (ASD) will participate in the study. The children with ASD will be recruited and tested at the clinical facilities of the Institute for Biomedical Research and Innovation of the National Research Council of Italy (IRIB-CNR) in Messina. To be included in the study the child needs to have an ASD diagnosis based on the Diagnostic and Statistical Manual, fifth edition (DSM-5) criteria from a licensed clinical child neuropsychiatrist but no established intellectual disability (ID) diagnosis.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Video analysis of performance | The video analysis needs approximately 15 minutes per child
  The videos of the interviews were analyzed by a single observer. For each child, the observer evaluated both the child's interactions, one with a person and another with the robot. The assessment included the child's attention, measured by the frequency and duration of the child's gazes towards the interaction partner. Additionally, the observer recorded the number of imitations of the partner's actions, limited to a maximum of four imitations. Finally, to evaluate repetitive and stereotyped behaviors, the observer counted the sequences of these behaviors and the number of repetitions within each sequence. A sequence was defined as a continuous repetition of the same behavior type, with pauses or interruptions considered as separate sequences. If the child paused and resumed the same or a different behavior, each restart was counted as a new sequence.

SECONDARY OUTCOMES:
Heart rate | The test needs approximately 30 minutes
  The polar sensor detects the electrical activity of the heart and calculates heart rate in beats per minute (bpm).Typically it is worn on the wrist or chest.
Heart rate variability | The test needs approximately 30 minutes
  The Polar sensor measures the time intervals between successive heart beats and calculates Heart Rate Variability (HRV) in milliseconds (ms). Typically it is worn on the wrist or chest.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costa AP, Charpiot L, Lera FR, Ziafati P, Nazarikhorram A, van der Torre L, Steffgen GA (2018) Comparison between a person and a robot in the attention, imitation, and repetitive and stereotypical behaviors of children with Autism Spectrum Disorder. In: Proceedings workshop on Social human-robot interaction of human-care service robots at HRI2018
- [Background] Zheng Z, Young EM, Swanson AR, Weitlauf AS, Warren ZE, Sarkar N. Robot-Mediated Imitation Skill Training for Children With Autism. IEEE Trans Neural Syst Rehabil Eng. 2016 Jun;24(6):682-91. doi: 10.1109/TNSRE.2015.2475724. Epub 2015 Sep 3. PMID 26353376
- [Background] Zorcec T, Ilijoski B, Simlesa S, Ackovska N, Rosandic M, Popcevic K, Robins B, Nitzan N, Cappel D, Blum R. Enriching Human-Robot Interaction with Mobile App in Interventions of Children with Autism Spectrum Disorder. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2021 Oct 26;42(2):51-59. doi: 10.2478/prilozi-2021-0021. PMID 34699714